CLINICAL TRIAL: NCT00651963
Title: Open Label Study Evaluating The Use Of Combination Therapy Of Ezetimibe And Statins In Patients With Dyslipidemia In Colombia
Brief Title: Open Label Study Evaluating The Use Of Combination Therapy Of Ezetimibe And Statins In Patients With Dyslipidemia In Colombia (0653-141)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0653-141; MK0653-141; 2008_007
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Lipid Metabolism Disorder
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — Ezetimibe

INTERVENTIONS:
Drug: ezetimibe — Ezetimibe 10 mg daily was added during 4 weeks.
  The patients continued taking their usual Statin without titrating the dose.
  Other Names: Zetia®; MK0653

SUMMARY:
Gather additional efficacy and safety (pharmacovigilance) information in the usual daily care in patients with Dyslipidemia on ezetimibe under real conditions in Colombia associated with statins.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Lipid Metabolic Disorder as Per ATP III who have not reached the goals and who are on statins for at least 4 weeks Or those who require LDL reductions Over 50% to reach the ATP III goals or who need statins in accordance their risk score

Exclusion Criteria:

* Pregnancy, Breast Feeding
* Moderate/Sever Liver Disease: Child Score > Or = To 7
* Fibrates Terminal Disease
* Contraindications To Receive ezetimibe
* Contraindications To Receive Statins
* Mental Disability
* Hypersensitivity To ezetimibe
* On another Clinical Research Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-09; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Lipid profile | Over 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC